CLINICAL TRIAL: NCT04506593
Title: Gastrointestinal Motility Diagnosis Registry
Brief Title: Indiana University Gastrointestinal Motility Diagnosis Registry
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John M. Wo, Douglas Rex Professor of Gastroenterology and Hepatology; Director of GI Motility and Neurogastroenterology Unit, Indiana University
Other Study IDs: GI Database; 1403899260 (Other: Indiana University IRB)
Record Dates: First submitted 2016-07-16; First posted 2020-08-10 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Eosinophilic Esophagitis; Gastroesophageal Reflux Disease (GERD); Gastroparesis; Functional Vomiting; Irritable Bowel Syndrome (IBS); Constipation; Chronic Intestinal Pseudo-obstruction; Fecal Incontinence; Small Intestinal Bacterial Overgrowth
Keywords: Eosinophilic esophagitis; Chronic intestinal pseudo-obstruction; Small Bowel dysmotility; SIBO; Vomiting; Functional dyspepsia; Functional bloating; Gastroparesis
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastroesophageal Reflux; Gastroparesis; Irritable Bowel Syndrome; Constipation; Fecal Incontinence; Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention

SUMMARY:
Develop a registry (list of patients) with accurate clinical motility diagnosis. This registry will help the doctors to identify the patients with specific disease conditions. It will also help in promoting future research in gastroenterology motility disorders

DETAILED DESCRIPTION:
Develop a registry (list of patients) of patients seen the clinics with motility disorders. Motility diagnosis based on billing diagnostic codes are not accurate. Motility diagnosis will be made by physicians with specialized in GI Motility, based on clinical consensus of diagnostic criteria. The information gathered from the database will be used to help promote future clinical research in the GI motility and Neurogastroenterology Unit at Indiana University School of Medicine.

Gastrointestinal motility symptoms are very common. It encompasses a wide range of problems, such as dysphagia, heartburn, nausea, emesis, food regurgitation, abdominal distension, weight loss, postprandial bloating, constipation, and diarrhea. An accurate diagnosis is essential in order to promote cost-effective treatment and future research to benefit patients with GI motility disorders

Specific Aims

1. Primary Aim: Identification of patients by accurate motility diagnosis
2. Secondary Aims:

   1. To develop Patient Reported Outcome (PRO) measurements in patients with small intestinal bacterial overgrowth (SIBO)
   2. To develop Patient Reported Outcome (PRO) measurements in patients with gastroparesis

ELIGIBILITY:
Inclusion Criteria:

1. Patients who presented to the GI outpatient clinics, in-patient consult service, and outpatient endoscopy centers within the Division of Gastroenterology and Hepatology
2. Carries a diagnosis of GI motility disorder based on the diagnostic criteria listed in table

Exclusion Criteria:

1. Coexisting medical conditions that may limiting participation in clinical research trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients who presented to the GI outpatient clinics, in-patient consult service, and outpatient endoscopy centers within the Division of Gastroenterology and Hepatology
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-11; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Identification of patients by accurate motility diagnosis | .through study completion, an average of 10 years
  Motility diagnosis will be made by physicians with specialized in GI Motility, based on consensus diagnostic criteria. The information gathered from the database will be used to help promote future clinical development and research in GI motility disorders.

SECONDARY OUTCOMES:
Patient Reported Outcome (PRO) Measurements in Patients with Small Intestinal Bacterial Overgrowth (SIBO) | through study completion, an average of 10 years
  SIBO-disease specific patient questionnaire will be compared between patients with aerodigestive tract SIBO and coliform SIBO
Patient Reported Outcome (PRO) Measurements in Patients with Gastroparesis | through study completion, an average of 10 years
  Patient Assessment of GI - Symptom (PAGI-SYM) scores will be compared between patients with emesis-predominant, dyspeptic-predominant, and regurgitation-predominant gastroparesis.

CONTACTS AND LOCATIONS:
Overall Officials: John m Wo, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
observational registry